CLINICAL TRIAL: NCT01998490
Title: Animal-assisted or Robot-assisted Interventions in Health Promotion for Elderly With Dementia: Impact on Factors Related to the Risk of Falls, on Evidence Based Practice and on the Relatives' Burden
Brief Title: Animal-assisted or Robot-assisted Interventions in Health Promotion for Elderly With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Life Sciences (Other)
Collaborators: Vestfold University College (Other)
Responsible Party: Principal Investigator, Camilla Ihlebæk, Professor, Norwegian University of Life Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012/1144
Record Dates: First submitted 2013-11-19; First posted 2013-11-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Animal-assisted activity (Experimental): 30 minutes group session with animal-assisted activity twice a week for 12 weeks in groups of 4-6 participants.
  Interventions: Other: Animal-assisted activity
- Robot-assisted activity (Experimental): 30 minutes group session with robot-assisted activity with the robot seal Paro twice a week for 12 weeks in groups of 4-6 participants
  Interventions: Other: Robot-assisted activity
- Control (No Intervention): Control group with treatment as usual

INTERVENTIONS:
Other: Animal-assisted activity
  Arms: Animal-assisted activity
Other: Robot-assisted activity
  Arms: Robot-assisted activity

SUMMARY:
The overall research aim of this study is to investigate changes in measures related to the risk of falls among elderly with dementia participating in animal-assisted or robot-assisted interventions. In addition the study will investigate how knowledge transfer occurs among involved health personnel, and how knowledge is refined and transformed as practical competence. The design will be a prospective and cluster randomized multicenter trial, but mixed-methods will be used to target different outcomes. The study population will be elderly (age above 65) at nursing homes diagnosed with dementia, or having a cognitive deficit. The intervention will consist of 30 minutes sessions with animal-assisted activity or robot-assisted activity two times a week for 12 weeks in groups of 4-6 participants. Control groups will receive treatment as usual. Research questions:

1. Is there an effect in use of ordinary and optional medication among elderly persons with dementia at nursing homes participating in animal-assisted or robot-assisted interventions compared to a control group?
2. Is there an effect on agitation, restlessness and depression among elderly persons with dementia at nursing homes participating in animal-assisted or robot-assisted interventions compared to a control group?
3. Is there an effect on social interaction, activeness and wellbeing among elderly persons with dementia at nursing homes participating in animal-assisted or robot-assisted interventions compared to a control group?

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of dementia or having a cognitive deficit measured as a score less than 25 on Mini-Mental State Examination.

Exclusion Criteria:

* Fear of dogs
* Dog allergy
* Need of wheel chair

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in Norwegian version of The Brief Agitation Rating Scale | Second last or last week before the intervention starts, after 4 and 8 weeks of the intervention, and first or second week after end of intervention. A follow-up measure 3 months after end of the intervention

OTHER OUTCOMES:
Change in Norwegian version of Cornell scale for depression | Second last or last week before the intervention starts, after 4 and 8 weeks of the intervention, and first or second week after end of intervention. A follow-up measure 3 months after end of the intervention
Change in Norwegian version of QUALID | Second last og last week before the intervention starts, after 6 weeks of the intervention, and first or second week after end of intervention. A follow-up measure 3 months after end of the intervention
Change in behaviours, engagement and well-being measured by use of Dementia Care Mapping | Second last or last week before the intervention starts, after 6 weeks of the intervention, and first or second week after end of intervention.
Change in physical activity measured by use of Actigraphy | Second last or last week before the intervention starts, after 6 weeks of the intervention, and first or second week after end of intervention
  A device worn by the participants for one week at each time point of measure, night and day, measuring physical movement.
Video recordings | After two and ten weeks of the interventions
  The video recorded will be analyzed with respect to social interaction and group dynamics
Change in use of ordinary and optional medication | Second last or last week before the intervention starts, first or second week after end of intervention and 3 months after end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Ihlebæk, PhD, Principal Investigator — Norwegian University of Life Sciences
Locations (15):
- Norway (15):
  - Pålsetunet bo- og servicesenter, Fet
  - Solliheimen Sykehjem, Fredrikstad
  - Solheimen senter, Halden
  - Frida Sykehjem, Larvik
  - Lørenskog Sykehjem, avd. Losbyveien, Lørenskog
  - Løreskog sykhjem, avd Krydderhagen, Lørenskog
  - Orkerød Sykehjem, Moss
  - Ryggeheimen, Moss
  - Gipø Sykehjem, Nøtterøy
  - Greverud Sykehjem, Oppegård
  - Høyås Sykehjem, Oppegård
  - Sandetun Sykehjem, Sande
  - Kamfjordhjemmet, Sandefjord
  - Sørvald bo- og behandlingssenter, Sørum
  - Tjøme Sykehjem, Tjøme

REFERENCES:
- [Derived] Joranson N, Pedersen I, Rokstad AM, Ihlebaek C. Change in quality of life in older people with dementia participating in Paro-activity: a cluster-randomized controlled trial. J Adv Nurs. 2016 Dec;72(12):3020-3033. doi: 10.1111/jan.13076. Epub 2016 Aug 16. PMID 27434512